CLINICAL TRIAL: NCT03529318
Title: Mucosal Innate Immune Activation in Chronic Intestinal Disorders
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 217718
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Irritable Bowel Syndrome; Inflammatory Bowel Diseases
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biopsies from endoscopy — 1) Patients scheduled for endoscopy (EGD or colonoscopy) for IBD will be consented to allow physicians who are performing endoscopies to take additional biopsies and blood samples for "research purposes".

SUMMARY:
Crohn's disease and ulcerative colitis are types of chronic intestinal disorder called inflammatory bowel diseases (IBD) that can affect the small and large bowel causing symptoms of abdominal pain, diarrhea, blood in the stool, and weight loss. Irritable bowel syndrome (IBS) is a milder form of IBD, with symptoms of abdominal pain, bloating, diarrhea or constipation, and blood in the stool. It is not known what causes diseases such as IBD and IBS. This study will look at the events in the gut that leads to leaky gut and inflammation in patients with IBD and IBS. The study will also see if medications such as rifaximin and mesalamine may reduce the amount of leaky gut.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-years old and older
* Presenting at the University of Arkansas for Medical Sciences (UAMS) Endoscopy center to undergo endoscopy with biopsy for surveillance, screening or diagnosis.

Exclusion Criteria:

* Subjects classified in an anesthesia risk group , American Society of Anesthesiologists Class (ASA) ≥ 4,
* history of bleeding diathesis or coagulopathy
* stroke or transient neurological attack within the last 6 months
* pregnancy
* currently on blood thinners (excepting aspirin)
* subject is unable to consent themselves

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population includes patients with known Crohn's disease, ulcerative colitis and indeterminant colitis. Patients will be recruited after they check in to the endoscopy unit, and before their endoscopic procedure, prior to any pre-procedure sedation medications having been given. All participants are undergoing endoscopy with biopsy for surveillance, screening, , diagnosis , or assessment of treatment. If no biopsy specimens are taken from subjects for diagnosis, no biopsy samples are taken for research purposes. The subject enrollment goal is 60 separate subjects with Crohn's disease, ulcerative colitis and indeterminant colitis or Irritable bowel syndrome. The subjects' participation will be limited to in the endoscopy suite.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Estimated)

PRIMARY OUTCOMES:
The number of specimens showing elevated levels of mucosal innate immune activation | Up to 2 years
  Determining the level of mucosal innate immune activation by staining, organoid culture, Western blot analysis, and cytokine expression on biopsy samples in IBD and IBS patient samples.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tharian, MD, Principal Investigator — University of Arkansas; Julia Liu, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No